CLINICAL TRIAL: NCT00585754
Title: Guanfacine to Reduce Stress-Induced Cocaine/Alcohol Craving and Relapse
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Yale University (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Principal Investigator, Rajita Sinha, Professor, Yale University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 0512000886; R01DA027130 (NIH)
Record Dates: First submitted 2007-12-22; First posted 2008-01-03 (Estimated); Last update posted 2016-11-30 (Estimated); Status verified 2016-11

CONDITIONS: Cocaine Dependent; Alcohol Dependent
MeSH Terms: interventions — Guanfacine

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Guanfacine (Active Comparator)
  Interventions: Drug: Guanfacine
- PLA (Placebo Comparator)
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Guanfacine — 1.5mg BID
  Arms: Guanfacine
Drug: Placebo — placebo
  Arms: PLA

SUMMARY:
This study aims to test the preliminary efficacy of 3.0 mg of guanfacine (GFC) daily versus placebo in cocaine and/or alcohol dependent individuals. This proposal is a laboratory and treatment outcome study to examine the effects of guanfacine on brief exposure to stress, drug cues and neutral situations on cocaine/alcohol craving, mood and neurobiological reactivity in a sample of cocaine and/or alcohol dependent individuals. Guanfacine will be beneficial for reduction in stress and drug cue induced craving and related arousal. In a sample of 60 cocaine and/or alcohol dependent men and women, we propose to examine (a) differences in measures of cocaine craving, emotion state, hypothalamic-pituitary-adrenal (HPA) activation, physiological arousal and plasma catecholamine response to stress imagery and to drug cue imagery as compared to neutral imagery; (b) reduction in cocaine/alcohol abstinence symptoms; and (c) improvement in cocaine and alcohol treatment outcomes as measured by increasing abstinence, reduction in cocaine/alcohol use and increased treatment attendance. Hypothesis 1: Guanfacine will decrease stress-induced cocaine craving, negative emotions and related arousal in the laboratory as compared to placebo. Hypothesis 2a: As compared to the PLA group, the GFC group will show significant reductions in protracted withdrawal symptoms as measured by the CSSA/CIWA during the 9-week treatment period.

Hypothesis 2b: As compared to the PLA group, a higher percentage of the GFC patients will remain abstinent during the 9-week treatment period with a higher percent of negative cocaine urines and alcohol-free days.

Hypothesis 2c: The GFC group will show greater adherence to treatment as measured by the days in treatment as compared to the Pla group.

ELIGIBILITY:
Inclusion Criteria:

* Male or female individuals, ages 18 and above, meeting current DSM-IV criteria for cocaine and/or alcohol dependence.
* COCAINE SAMPLE: meet current DSM-IV criteria for cocaine dependence; documented positive urine toxicology screen for cocaine at intake
* ALCOHOLIC SAMPLE: meet current DSM-IV criteria for alcohol dependence
* Subject has voluntarily given informed consent and signed the informed consent document.
* Able to read English and complete study evaluations.

Exclusion Criteria:

* Meet current criteria for dependence on another psychoactive substance, excluding nicotine and caffeine;
* Any current use of opiates or past history of opiate abuse/dependence;
* Current use of any psychoactive drugs, including anxiolytics, antidepressants, naltrexone or antabuse;
* Any psychotic disorder or current Axis I psychiatric symptoms requiring specific attention, including need for psychiatric medications for current major depression and anxiety disorders
* Significant underlying medical conditions such as cerebral, renal, thyroid or cardiac pathology which in the opinion of study physician would preclude patient from fully cooperating or be of potential harm during the course of the study;
* Abstinent from cocaine for more than two weeks prior to admission.
* Hypotensive individuals with sitting blood pressure below 90/50 mmHG.

Ages: 18 Years to 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 75 (Actual)
Dates: Start 2006-04; Primary Completion 2016-06 (Actual); Study Completion 2016-06 (Actual)

PRIMARY OUTCOMES:
stress-induced cocaine craving and negative emotions | 5 years

SECONDARY OUTCOMES:
Drug and alcohol use | over ninety days

CONTACTS AND LOCATIONS:
Overall Officials: Rajita Sinha, PhD, Principal Investigator — Yale University
Locations (1):
- Yale University School of Medicine: Yale Stress Center, New Haven, Connecticut, United States

REFERENCES:
- [Derived] Milivojevic V, Fox HC, Jayaram-Lindstrom N, Hermes G, Sinha R. Sex differences in guanfacine effects on stress-induced stroop performance in cocaine dependence. Drug Alcohol Depend. 2017 Oct 1;179:275-279. doi: 10.1016/j.drugalcdep.2017.07.017. Epub 2017 Aug 10. PMID 28823835
- [Derived] Fox HC, Morgan PT, Sinha R. Sex differences in guanfacine effects on drug craving and stress arousal in cocaine-dependent individuals. Neuropsychopharmacology. 2014 May;39(6):1527-37. doi: 10.1038/npp.2014.1. Epub 2014 Jan 7. PMID 24395021